CLINICAL TRIAL: NCT00801151
Title: A Phase I Clinical Trial of Vorinostat in Combination With Vinorelbine in Patients With Advanced Cancer.
Brief Title: Vorinostat in Combination With Vinorelbine in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr Jean-Pierre DELORD, Institut Claudius REGAUD
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07 GENE 05; NCT00801840 (obsolete NCT alias)
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-05

CONDITIONS: Malignant Solid Tumour
MeSH Terms: interventions — Vorinostat; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat, vinorelbine (Experimental): Vorinostat will be administered orally at the starting dose of 200 mg po qd 7/21(weekly schedule) in combination with the standard dose of vinorelbine 25mg/m² per week as intravenous infusion over 10 minutes starting 4 hours after vorinostat administration.
  Interventions: Drug: Zolinza (vorinostat), vinorelbine

INTERVENTIONS:
Drug: Zolinza (vorinostat), vinorelbine — Vorinostat will be administered orally at the starting dose of 200 mg po qd 7/21(weekly schedule) in combination with the standard dose of vinorelbine 25mg/m² per week as intravenous infusion over 10 minutes starting 4 hours after vorinostat administration.
  Barring dose limiting toxicities the dose of vorinostat will escalate in several steps (300 mg po qd 7/21 days, 300 mg po qd 21/21 days, 400 mg po qd 7/21 days, 400 mg po qd 21/21 days).
  Patients may receive a maximum of 6 cycles of study medication.
  Other Names: Vorinostat, MK 0683, SAHA

SUMMARY:
This is a multi-center, open-label non-randomized dose-escalation trial of vorinostat given in combination with vinorelbine. Cohorts will be treated with a fixed dose of vinorelbine (25mg/m²/week continuously, representing the schedule that has been approved). Patients eligible will be enrolled into a standard 3+3 design with a starting dose of vorinostat at 200 mg po qd 7/21 (weekly schedule). Then, further dose levels will be explored. Toxicity of the schedule will be assessed during the first cycle. Patients may receive up to 6 cycles of study medication. Blood samples will be collected at specified time points to assess pharmacokinetic endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically-confirmed metastatic or locally advanced cancer.
* Patient is ≥ 18 years of age on day of signing informed consent.
* Patient must have performance status < 1 on the ECOG performance scale.
* Patient must have adequate organ function as indicated by the following laboratory values:

  * Hematological: absolute neutrophil count (ANC) ≥ 1,5x109/L; platelets ≥ 100 x109/L; hemoglobin ≥ 9 g/dL
  * Renal : calculated creatinine clearance b ≥ 60 mL/min
  * Hepatic : serum total bilirubin ≤ 1.5 X ULN ; AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN; alkaline phosphatase if > 2.5 X ULN, then liver fraction should be ≤ 2.5 X ULN
  * Coagulation : prothrombin time (PT) ≤1.2 X ULN ; partial thromboplastin time (PTT) ≤1.2 X ULN

    1. Patients should have adequate bone marrow function without the current use of colony stimulating factors
    2. Creatinine clearance should be calculated according to Cockcroft-Gault formula
* For female patients of childbearing potential: must have a negative serum pregnancy test within 72 h before drug administration
* Male and Female patients of childbearing potential must agree to use an adequate method of contraception throughout the study starting with Visit 1 and for at least 30 days after the last dose of study medication.
* Patient has voluntarily agreed to participate by giving written informed consent.
* Patient must be available for periodic blood sampling, study related assessments, and management at the treating institution of the duration of the study.

Exclusion Criteria:

* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent.
* Patient pre-treated with one of the two investigational compounds (ie; vinorelbine or vorinostat)
* Patients with active CNS metastases and/or carcinomatous meningitis and uncontrolled brain metastases are excluded. However, patients with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for 3 months prior to entry as defined as: (1) no evidence of new or enlarging CNS metastasis (2) off steroids or on a stable dose of steroids.
* Patient has known hypersensitivity to the components of study drug or its analogs.
* Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse.
* Patient is pregnant or nursing,
* Patient is known to be Human Immunodeficiency Virus (HIV)-positive.
* Patient has known history of Hepatitis B or C.
* Patient with a history of a prior malignancy with the exception of cervical intraepithelial neoplasia; basal cell carcinoma of the skin; adequately treated localized prostate carcinoma with PSA <1.0; or who has undergone potentially curative therapy with no evidence of that disease for five years, and who is deemed at low risk for recurrence by his/her treating physician
* Patient has preexisting grade 2 or higher neuropathy
* Patients who had received radiotherapy to more than 30% of the bone marrow surface (i.e whole pelvis)
* Patients under law protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of vorinostat administered in combination with standard doses of vinorelbine. | at the end of the trial

SECONDARY OUTCOMES:
To assess the pharmacokinetics of vorinostat and vinorelbine when administered in combination. | at the end of the trial
To assess the safety and tolerability of this regimen in advanced solid tumors. | at the end of the study
To make a preliminary assessment of the efficacy of the combination, in terms of response rate, response duration, time to response and time to progression. | At the end of the trial
To evaluate predictive pharmacodynamic biomarkers (e.g., histone acetylation in peripheral blood) when vorinostat is administered in combination with vinorelbine. | At the end of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Delord, MD, PhD, Principal Investigator — Institut Claudius Regaud
Locations (3):
- France (3):
  - Centre René GAUDUCHEAU, Nantes Saint Herblain
  - Institut Curie, Paris
  - Institut Claudius REGAUD, Toulouse